CLINICAL TRIAL: NCT01519375
Title: Cross-sectional, Observational Real Life Study on NSAIDs Treated Patients With Osteoarthritis, Rheumatoid Arthritis and Ankylosing Spondylitis: Assessment of Patient Adherence to PPI Treatment
Brief Title: Assessment of NSAID-treated Patients Adherence to Co-prescribed Proton Pump Inhibitor (PPI)
Acronym: CONVOY
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RSE-ATC-2011/1
Record Dates: First submitted 2012-01-23; First posted 2012-01-26 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Ankylosing Spondylitis
Keywords: Osteoarthritis; Rheumatoid Arthritis; Ankylosing Spondylitis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with Osteoarthritis, Rheumatoid Arthritis and Ankylosing Spondylitis, 18 years or older

SUMMARY:
The primary objective of this cross-sectional observational real life study is to investigate the patient reported adherence to PPI, when prescribed as prevention of NSAID associated GI Ulcers to patients prescribed a NSAID. Patients included have Osteoarthritis, Rheumatoid Arthritis or Ankylosing Spondylitis. Adherence will be assessed by patient questionnaires.

DETAILED DESCRIPTION:
Cross-sectional, observational Real Life study on NSAIDs treated patients with Osteoarthritis, Rheumatoid Arthritis and Ankylosing Spondylitis: Assessment of patient adherence to PPI treatment

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis (documented in the medical record) of OA, RA or AS
* Prescription of oral NSAID treatment for OA, RA or AS, where low dose is not sufficient
* Prescription of PPI for prevention of NSAID associated GI ulcers, with instruction to take PPI same day as when taking NSAID.

Exclusion Criteria:

* Participating in any clinical trial involving PPI or NSAID
* Patients prescribed PPI as acute treatment of GI events or symptoms within 8 weeks
* Inability to complete PROs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 100 patients having Osteoarthritis (OA), Rheumatoid Arthritis (RA) and Ankylosing Spondylitis (AS) selected from medical records at involved clinics. The investigator will select the patients in order of date by latest visits to the clinic and backwards. The patients will be selected from 4-6 involved primary care and and specialist clinics.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Patient reported adherence to PPI treatment on actual days of NSAID treatment. | 7 days

SECONDARY OUTCOMES:
Proportion of patients with reported adherence ≤ 80%. | 7 days
Patient adherence to prescribed ASA treatment. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Stratelis, MD, PhD, Study Director — AstraZeneca Nordics, B674:4 151 87 Södertälje, Sweden; Kenneth Henriksson, MD, Principal Investigator — Reuma City, 111 52 Stockholm, Sweden
Locations (8):
- Sweden (8):
  - Research Site, Kristianstad
  - Research Site, Kristinehamn
  - Research Site, Limhamn
  - Research Site, Partille
  - Research Site, Skanör
  - Research Site, Stockholm
  - Research Site, Ullanger
  - Research Site, Vännäs